CLINICAL TRIAL: NCT02444780
Title: Observational Study on Plasma Glutamine Levels Before and After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Other Study IDs: nWMO 115
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Glutamin Level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elective cardiac surgery patients: consecutive patients who undergo elective cardio-thoracic surgery during a 6 to 8 week period
  Interventions: Procedure: no intervention, blood is sampled for routine

INTERVENTIONS:
Procedure: no intervention, blood is sampled for routine — no intervention, blood sampled for standard evaluation will be used for determination of plasma glutamin

SUMMARY:
Earlier studies showed that a low glutamine level at acute admission on the ICU is associated with a poor outcome [3,4]. Recently, we found that a low plasma glutamine is correlated with severity of illness and presence of an infection after non-elective ICU admission [5, submitted].

DETAILED DESCRIPTION:
It is known that major surgery induces a stress response characterised by hormonal release and inflammatory processes [6,7]. This surgical stress response resembles the catabolic stress which is found in other forms of critical illness. We did not measure plasma glutamine before surgery so it is unknown whether the plasma glutamine level was already low before surgery in these patients or that the lowering of plasma glutamine level is a consequence of surgery. Most of the patients in the elective surgery group in our study underwent cardiac surgery with use of cardiopulmonary bypass; it is known that extracorporeal circulation induces an inflammatory response but there are no clinical data on the effects on plasma glutamine or on post-operative course in relation to plasma glutamine levels [8,9].

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective cardiac surgery

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who undergo elective cardio-thoracic surgery during a 6 to 8 week period.
  We aim to include at least 90 patients.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
plasma glutamine | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Buter, MD, Principal Investigator — MCL

REFERENCES:
- [Derived] Buter H, Koopmans M, Kemperman R, Jekel L, Boerma C. Plasma glutamine levels before cardiac surgery are related to post-surgery infections; an observational study. J Cardiothorac Surg. 2016 Nov 25;11(1):155. doi: 10.1186/s13019-016-0549-1. PMID 27884211